CLINICAL TRIAL: NCT06625307
Title: A First-in-human Randomised, Placebo-controlled and Double-blinded Single Ascending Dose Study Investigating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Administrations of NNC0537-1482 in Healthy Participants.
Brief Title: A Research Study on the Effects of NNC0537-1482 in Healthy Individuals When Injected Under the Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6537-7650; U1111-1298-6922 (Other: World Health Organization (WHO)); 2024-514431-18 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- NNC0537-1482 Dose level 1 (Experimental): Participants will be administered a single dose of dose level 1 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482; Drug: Placebo
- NNC0537-1482 Dose level 2 (Experimental): Participants will be administered a single dose of dose level 2 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482; Drug: Placebo
- NNC0537-1482 Dose level 3 (Experimental): Participants will be administered a single dose of dose level 3 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482; Drug: Placebo
- NNC0537-1482 Dose level 4 (Experimental): Participants will be administered a single dose of dose level 4 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482; Drug: Placebo
- NNC0537-1482 Dose level 5 (Experimental): Participants will be administered a single dose of dose level 5 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482; Drug: Placebo
- NNC0537-1482 Dose level 6 (Experimental): Participants will be administered a single dose of dose level 6 of NNC0537-1482 subcutaneously.
  Interventions: Drug: NNC0537-1482; Drug: Placebo
- Placebo (Placebo Comparator): Participants will be administered a single dose of Placebo matched to NNC0537-1482 subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0537-1482 — Administered via subcutaneous route
  Arms: NNC0537-1482 Dose level 1; NNC0537-1482 Dose level 2; NNC0537-1482 Dose level 3; NNC0537-1482 Dose level 4; NNC0537-1482 Dose level 5; NNC0537-1482 Dose level 6
Drug: Placebo — Administered via subcutaneous route

SUMMARY:
The study is testing a new medicine to potentially treat people with heart failure. The main purpose of the study is to see if the new study medicine is safe and how it works in the body. It is the first time NNC0537-1482 (the new study medicine) is tested in humans and will be tested in healthy individuals (men and postmenopausal women). Participant will either get NNC0537-1482 or placebo (a "dummy medicine" without any active ingredients). Which treatment the participant get is decided by chance and the participant will only get either the study medicine or placebo on one occasion. It will be injected under the skin of the stomach by the study staff and the number of injections will depend on the cohort participant is assigned to. NNC0537-1482 cannot be prescribed by doctors. The study consists of 6 cohorts (groups) with 6 different dosing levels. The study will last for about 9 months. Participation in the study will last up to 42 days (depending on the cohort participant are assigned to) with an additional screening period that can be up to 28 days. Participant will have up to 10 visits to the clinic during the study period. However, the total number of visits depend on which cohort participant is assigned to.

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal female.
* Age 22-55 years (both inclusive) at the time of signing the informed consent.
* Body Mass Index (BMI) between 18.5 and 30.0 kilogram/meter per square (kg/m^2) (both inclusive) at screening.
* Considered eligible and generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Use of prescription or non-prescription medicinal products, including herbal medications, within 14 days before screening. Occasional use of over-the-counter vitamins, or paracetamol or Non-steroidal anti-inflammatory drugs (NSAIDs) at their labelled doses for mild pain is permitted.
* Any condition which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Orthostatic hypotension, defined as a decrease in systolic blood pressure greater than or equal to 20 millimetres of mercury (mmHg) or a decrease in diastolic blood pressure greater than or equal to 10 (mmHg) from supine to standing after 3 minutes, at the screening visit.
* Any laboratory safety parameters at screening outside the below laboratory ranges for:

  * Alanine Aminotransferase (ALT) greater than (>) Upper normal limits (UNL) plus (+) 10 Percentage (%)
  * Aspartate Aminotransferase (AST) > Upper limit normal (ULN) +20%
  * Bilirubin > ULN + 20%
  * Creatinine > ULN + 10%

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2025-05-04 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAE) in cohorts 1 and 2 | From pre-dose on Day 1 until completion of the End of study visit (V10) at Day 15
  Number of events.
Number of treatment emergent adverse events (TEAE) in cohort 3 | From pre-dose on Day 1 until completion of the End of study visit (V10) at Day 22
  Number of events.
Number of treatment emergent adverse events (TEAE) in cohorts 4, 5 and 6 | From pre-dose on Day 1 until completion of the End of study visit (V10) at Day 40
  Number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency '(dept. 2834)', Study Director — Novo Nordisk A/S
Locations (1):
- ICON - location Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: https://novonordisk-trials.com